CLINICAL TRIAL: NCT03153475
Title: Multi-Center Clinical Evaluation of the ATTUNE® Revision System in Revision Total Knee Arthroplasty
Brief Title: ATTUNE Revision System in the Revision Total Knee Arthroplasty Population
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSJ-2016-02
Record Dates: First submitted 2017-05-07; First posted 2017-05-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Revision Total Knee Arthroplasty
Keywords: Revision knee surgery, implant replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ATTUNE Revision Knee System (Other): The ATTUNE Revision system is complementary to the ATTUNE primary knee portfolio and includes both rotating platform (RP) and fixed bearing (FB) configurations. The system includes a full compliment of implants designed to address the challenges faced in revision knee surgeries. These implants include Stemmable tibial and femoral components, augments, sleeves and offsets
  Interventions: Device: ATTUNE Revision Knee System in Revision Total Knee Arthroplasty

INTERVENTIONS:
Device: ATTUNE Revision Knee System in Revision Total Knee Arthroplasty — Implants from the ATTUNE Revision Knee System will be used to treat subjects whose surgeons have determined their existing implants need to be removed and replaced.
  Other Names: previous unsuccessful knee replacement, knee revision

SUMMARY:
Five-year, Prospective, multi-center, non-randomized, non-controlled study of the ATTUNE® Revision total knee prostheses, utilizing the fixed bearing (FB) and rotating platform (RP) tibial component with the posterior stabilizing (PS) femoral component in revision total knee arthroplasty.

DETAILED DESCRIPTION:
The study is designed as a non-comparative, worldwide, multi-center study with up to 30 sites that will intend to implant a total of 400 Subjects (200 PS RP and 200 PS FB) with the study devices. The follow-up period of 5 years was selected to cover both the early post-operative period as well as the medium term period which is a good indicator of longer term survivorship.

The primary endpoint of survivorship at 5 years was selected to capture the time period during which the majority of revision failures occur while providing a good indication of long term survivorship. The secondary outcomes include commonly used measures of clinical performance that will allow for comparison with published literature. Additionally, patient reported outcomes, AORI bone defect classification , satisfaction and pain scores will be collected and analyzed.

Male and female Subjects, age 22-80 years, inclusive, with a failed primary knee arthroplasty, including unicompartmental or failed previous revision TKA, who are suitable candidates for revision TKA using the ATTUNE® Revision system are eligible for enrollment in this study. The use of the ATTUNE Revision system includes both partial and complete revision surgical procedures, including implantation of revision components as the second stage within a two-stage treatment for infection.

ELIGIBILITY:
Inclusion Criteria

1. Subject is male or female and between the ages of 22 and 80 years at the time of consent, inclusive.
2. Subject presents with a primary knee arthroplasty (primary TKA, unicompartmental) or prior revision TKA that requires a revision procedure of implanted tibial and/or femoral components.
3. The decision to perform a knee revision with the study device is regardless of the research.
4. Subject that is willing to give voluntary, written informed consent to participate in this clinical investigation and authorize the transfer of his/her information to the Sponsor
5. Subject is currently not bedridden
6. The devices are to be used according to the approved indications.Subject is able to read, and comprehend the Informed Consent Document as well as complete the required PROMs in either English or one of the available translations.

Exclusion Criteria:

1. The Subject is a woman who is pregnant or lactating.
2. Contralateral knee has already been enrolled in this study.
3. Subject had a contralateral amputation.
4. Subject is currently diagnosed with radicular pain from the spine that radiates into the limb to receive RTKA.
5. Subject has participated in a clinical investigation with an investigational product (drug or device) in the last three (3) months.
6. Subject is currently involved in any personal injury litigation, medical-legal or worker's compensation claims.
7. Subject, in the opinion of the Investigator, is a drug or alcohol abuser (in the last 5 years) or has a psychological disorder that could affect his/her ability to complete patient reported questionnaires or be compliant with follow-up requirements.
8. Subject was diagnosed and is taking prescription medications to treat a muscular disorder that limits mobility due to severe stiffness and pain such as fibromyalgia or polymyalgia.
9. Subject has a significant neurological or musculoskeletal disorder(s) or disease that may adversely affect gait or weight bearing activities (e.g., muscular dystrophy, multiple sclerosis, Charcot disease).
10. Subject has a medical condition with less than five (5) years life expectancy as determined by the Investigator.
11. Uncontrolled gout

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Survivorship | 5 Years
  To evaluate the 5 year survivorship using Kaplan-Meier survival analysis, with revision for any reason as the endpoint, for the ATTUNE® Revision TKA PS FB and PS RP configurations.

SECONDARY OUTCOMES:
Patient's Knee Implant Performance (PKIP) | Baseline, 2 and 5 yr timepoints
  Evaluate change from preoperative baseline to 2 and 5 yr timepoints in functional outcomes, satisfaction and quality of life assessments, as measured using the PKIP patient reported outcome measure (overalll and subscores)
Knee Injury and Osteoarthritis Outcome Score Short form (KOOS-PS) | Baseline, 2 year and 5 Year
  Evaluate change from preoperative baseline to 2 and 5 yr timepoints in functional outcomes assessments, as measured using the KOOS-PS patient reported outcome measures
American Knee Society Score | Baseline, 2 year, 5 year
  Evaluate change from preoperative baseline to 2 and 5 yr timepoints in functional outcomes assessments, patient satisfaction and expectations and clinical evaluations as measured using the AKS measure
EQ-5D-5L | Baseline, 2 year and 5 year
  Evaluate change from preoperative baseline to 2 and 5 yr timepoints in functional outcomes assessments, as measured using the EQ-5D-5L patient reported outcome measures
VAS Pain Score | Baseline, 2 year and 5 year
  Evaluate change from preoperative baseline to 2 and 5 yr timepoints in patient reported pain severity as measured using a modified VAS Pain Score (discrete numbers rather than a continual scale).
Patient Satisfaction | Baseline, 2 year and 5 year
  Evaluate change from preoperative baseline to 2 and 5 yr timepoints in patient reported satisfaction as measured using a Likert scale.
Adverse Events | Intraoperative, 6 weeks, 1 yr, 2 yrs., 3 yrs., 4 yrs., 5 yrs.
  Evaluate type and frequency of Adverse Events
Readmissions | 6 weeks, 1 yr, 2 yrs., 3 yrs., 4 yrs., 5 yrs
  Evaluate the timing, duration and reason for any readmissions stratified by adverse event type (operative site vs. systemic).
Survivorship | 1, 2, 3 and 4 years
  Evaluate survivorship of the ATTUNE® Revision TKA system for the PS FB and PS RP configurations and the combined PS FB and PS RP configurations using Kaplan-Meier survival analysis at 1, 2, 3, and 4 years.
Frequency of radiolucent line occurrence | 1, 2 and 5 years
  Evaluate ATTUNE® Revision TKA fixation through zonal radiographic analysis of the bone-implant interface at 1, 2 and 5 years after surgery compared to the first postoperative radiographs.
Anatomic Tibiofemoral Alignment | 1, 2 and 5 years
  Evaluate any changes in anatomic tibiofemoral alignment at 1, 2 and 5 yrs compared to the first postoperative radiographs.
femoral component alignment | 1, 2 and 5 years
  Evaluate any changes in femoral component alignment at 1, 2 and 5 yrs compared to the first postoperative radiographs.
Tibial component alignment | 1, 2 and 5 years
  Evaluate any changes in tibial component alignment at 1, 2 and 5 yrs compared to the first postoperative radiographs.
Restoration of joint line | First post-operative radiograph (1 day)
  Radiographically evaluate the restoration of joint line using the first postoperative radiographs according to the methodology of Figgie.

CONTACTS AND LOCATIONS:
Overall Officials: Sukhjeet Kaur, Study Director — Sponsor GmbH
Locations (38):
- United States (16):
  - Scripps Clinic Torrey Pines, San Diego, California
  - Colorado Joint Replacement, Denver, Colorado
  - Orthopaedic Center of the Rockies, Fort Collins, Colorado
  - Orthopedic Partners, Niantic, Connecticut
  - Florida Orthopedic Associates, DeLand, Florida
  - Arthroplasty Foundation, Louisville, Kentucky
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mery Hospital, Ozark, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Rothman Institute, Egg Harbor, New Jersey
  - UNC Orthopaedics, Chapel Hill, North Carolina
  - OrthoCarolina Hip and Knee Center, Charlotte, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Southern Joint Replacement Institute, Nashville, Tennessee
  - Texas Institute for Hip & Knee Surgery, Austin, Texas
  - Fondren Orthopedic Group, Houston, Texas
- Australia (2):
  - The Gold Coast Centre for Bone and Joint Surgery, Gold Coast
  - St. John of God Murdoch Hospital, Perth
- Krankenhaus der Barmherzigen Schwestern Linz Betriebsgesellschaft m.b.H., Linz, Austria
- MoRe Foundation, Antwerp, Belgium
- Canada (2):
  - London Health Sciences Centre University Hospital, London, Ontario
  - Concordia Joint Replacement, Winnipeg
- France (2):
  - CHRU La Cavale Blanche, Brest
  - Centre Hospitalier Universitaire de Rennes, Rennes
- Germany (2):
  - Klinik und Poliklinik für Orthopädie und Sportorthopädie am Klinikum rechts der Isar der Technischen Universität Münche, Munich
  - Asklepios Orthopädische Klinik Lindenlohe, Schwandorf in Bayern
- South Infirmary Public Hospital, Cork, Ireland
- CLINICHE GAVAZZENI SPA aka Humanitas Castelli, Bergamo, Italy
- University Hospital Maastricht, Maastricht, Netherlands
- Wellington Hospital, Wellington, New Zealand
- Kantonsspital Baselland (Bruderholz, Liestal, Laufen), Department of Orthopaedic Surgery and Traumatology, Basel, Switzerland
- United Kingdom (7):
  - Hampshire Hospitals NHS Foundation Trust, Basingstoke
  - Victoria Hospital NHS Fife, Kirkcaldy
  - Chapel Allerton Orthopaedic Centre, Leeds
  - James Cook University Hospital, North Yorks
  - The Robert Jones and Agnes Hunt Orthopaedic Hospital NHS Foundation Trust, Oswestry
  - Nuffield Orthopaedic Centre, Oxford
  - Wrightington Hospital, Wigan

IPD SHARING:
Plan to Share IPD: No